CLINICAL TRIAL: NCT06257251
Title: Silicone Particles in Breast Implant Capsules: a Retrospective Monocentric Study Evaluation of Silicone Bleeding
Brief Title: Silicone Particles in Breast Implant Capsules
Status: Recruiting | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Socorro ORTIZ, Head of plastic surgery departement, Brugmann University Hospital
Other Study IDs: CHUB-silicone
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Breast Implant Leakage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Histological slides of the capsule samples taken during breast implant capsulectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast implant capsulectomy: Patients admitted and operated at CHU-Brugmann hospital for surgical revision of their breast implants.
  Interventions: Other: Histological slides digitization

INTERVENTIONS:
Other: Histological slides digitization — Histological slides of the capsule samples taken during surgery will be collected for analysis and digitized. Using the NDPview2 software, the investigators will manually count the silicone particles present in the peri-prosthetic capsule and measure the surface area of the capsule to estimate the silicone particle density.

SUMMARY:
Breast implantation is one of the most common surgical procedures in plastic surgery. It is used to reconstruct a breast after mastectomy following cancer or to increase breast volume for aesthetic purposes. Since their introduction in the 1960s, silicone breast implants have been the subject of multiple controversies, and their safety has long been questioned. One of the initial concerns was silicone bleeding, which refers to the sweating of silicone gel through the implant's shell. Once outside the implant, silicone particles accumulate in the peri-prosthetic capsule, but they can also migrate to distant sites through the lymphatic system. These particles are not entirely biologically inert, as they initiate a foreign body inflammatory reaction characterized by the presence of macrophages and giant cells that cluster around the particles. The resulting chronic inflammation can be the source of local complications, such as granuloma formation or the onset of breast pain.

Silicone bleeding was first described in the 1970s and was particularly common with second-generation implants (1970-1982), which had thin shells and low-viscosity gel. Despite the technical improvements made to current breast implants, silicone can still be detected in the peri-prosthetic capsules of silicone breast implants. Most patients are asymptomatic, but they may occasionally experience local pain.

An increasing number of patients with breast implants are suffering for breast implant illness (BII) : a disease with nonspecific systemic signs and symptoms such as fatigue, skin rash, or headaches…etc, the precise etiology of which remains unexplained. Although the causative link has never been proven, some authors hypothesize that silicone could be responsible for these systemic complaints. While there is ongoing debate and research on the topic, some people believe that silicone bleeding from breast implants may contribute to the development of BII symptoms. However, it's important to note that the connection between silicone bleeding and BII has not been definitively proven.

It is a single center retrospective study that will include a total of 65 patients who have undergone breast implant capsulectomy. Capsulectomy is a surgical procedure involving the partial or complete removal of the peri-prosthetic capsule that forms around a breast implant. The peri-prosthetic capsule is a naturally occurring fibrous tissue that forms in response to the presence of the implant in the body. Sometimes, this capsule can become thickened, contracted, or cause complications such as capsular contracture, asymmetry, or pain. Capsulectomy can be performed as part of a surgical revision of breast implants to address these complications or for other reasons.

The main objective of this study is to quantify silicone particles in the periprosthetic capsules of breast implants using an innovative method of quantification based on histological examination of capsule specimens. The secondary objective is to compare the amount of silicone in capsules from different types of breast implants (saline or silicone) to assess whether texture, shell, silicone gel and time of implantation could influence silicone bleeding and breast implant illness.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted and operated at CHU-Brugmann Hospital (Horta & Brien)
* Surgery between January 2013 and October 2023
* Type of surgery: surgical revision of their breast implants requiring partial or complete sampling of the peri-prosthetic capsule.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted and operated at CHU-Brugmann (Horta & Brien) between January 2013 and October 2023 for surgical revision of their breast implants, requiring partial or complete sampling of the peri-prosthetic capsule.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Silicone particles quantity | 1 day
  Manual count of the silicone particles present in the peri-prosthetic capsule
Peri-prosthetic capsule thickness | 1 day
  Peri-prosthetic capsule thickness
Silicone particle's' size | 1 day
  Size of the silicone particles present in the peri-prosthetic capsule

CONTACTS AND LOCATIONS:
Overall Officials: Socorro Ortiz, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No